CLINICAL TRIAL: NCT00217373
Title: A Phase I Study of Sequential Vaccinations With Fowlpox-CEA(6D)-Tricom (B7.1/ICAM/LFA3) and Vaccinia-CEA (6D)-Tricom, in Combination With GM-CSF and Interferon-Alfa-2B in Patients With CEA-Expressing Carcinomas
Brief Title: Vaccine Therapy, GM-CSF, and Interferon Alfa-2b in Treating Patients With Locally Advanced or Metastatic Cancer That Expresses Carcinoembryonic Antigen (CEA)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2011-01347; NCI-2011-01347 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); NCI-5633; OSU-2005H0005; CDR0000439532; OSU 0312 (Other: Ohio State University Comprehensive Cancer Center); 5633 (Other: CTEP); P30CA016058 (NIH); U01CA076576 (NIH)
Record Dates: First submitted 2005-09-20; First posted 2005-09-22 (Estimated); Last update posted 2015-04-20 (Estimated); Status verified 2014-12

CONDITIONS: Adult Solid Neoplasm
MeSH Terms: interventions — Introns; Interferon alpha-2; sargramostim; Colony-Stimulating Factors

ARMS (1):
- Arm I (Experimental): COURSE I: Patients receive recombinant vaccinia-CEA(6D)-TRICOM vaccine SC on day 1. Patients also receive sargramostim (GM-CSF) SC on days 1-4 and IFN-α-2b* SC on days 9, 11, and 13.
  COURSES II-IV: Patients receive recombinant fowlpox-CEA(6D)-TRICOM vaccine SC on day 1. Patients also receive GM-CSF as in course 1 and IFN-α-2b* SC on days 1, 3, and 5.
  NOTE: *The initial cohort of 6 patients does not receive IFN-α-2b.
  Treatment repeats every 28 days for 4 courses in the absence of disease progression or unacceptable toxicity. After 4 courses, patients who do not have progressive disease or unacceptable toxicity may receive recombinant fowlpox-CEA (6D)-TRICOM vaccine, GM-CSF, and IFN-α-2b every 28 days for 2 more courses and then every 3 months for up to 2 years.
  Interventions: Biological: Recombinant Fowlpox-CEA(6D)/TRICOM Vaccine; Biological: Recombinant Interferon Alfa-2b; Biological: Recombinant Vaccinia-CEA(6D)-TRICOM Vaccine; Biological: Sargramostim

INTERVENTIONS:
Biological: Recombinant Fowlpox-CEA(6D)/TRICOM Vaccine — Given SC
  Other Names: fowlpox-CEA-B7.1/ICAM-1/LFA-3; Recombinant Fowlpox-CEA-TRICOM Vaccine; rF-CEA(6D)TRICOM
Biological: Recombinant Interferon Alfa-2b — Given SC
  Other Names: Alfatronol; Glucoferon; Heberon Alfa; IFN alpha-2B; Interferon alfa 2b; INTERFERON ALFA-2B; Interferon Alpha-2b; Intron A; Sch 30500; Urifron; Viraferon
Biological: Recombinant Vaccinia-CEA(6D)-TRICOM Vaccine — Given SC
  Other Names: rV-CEA(6D)-TRICOM; Vaccinia-CEA-TRICOM Vaccine
Biological: Sargramostim — Given SC
  Other Names: 23-L-Leucinecolony-Stimulating Factor 2; DRG-0012; Leukine; Prokine; rhu GM-CFS; Sagramostim; Sargramostatin

SUMMARY:
This phase I trial is studying the side effects and best dose of interferon alfa-2b when given together with vaccine therapy and GM-CSF in treating patients with locally advanced or metastatic cancer that makes CEA. Vaccines made from a gene-modified virus may help the body build an effective immune response to kill cancer cells that make carcinoembryonic antigen (CEA). Biological therapies, such as GM-CSF, may stimulate the immune system in different ways and stop cancer cells from growing. Interferon alfa-2b may interfere with the growth of cancer cells and slow cancer growth. Giving vaccine therapy together with GM-CSF and interferon alfa-2b may kill more cancer cells that make CEA.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the maximum tolerated dose and recommended phase II dose of interferon alfa-2b (IFN-α-2b) when administered with recombinant vaccinia-CEA(6D)-TRICOM vaccine, recombinant fowlpox-CEA(6D)-TRICOM vaccine, and sargramostim (GM-CSF) in patients with locally advanced or metastatic carcinoembryonic antigen (CEA)-expressing carcinoma.

SECONDARY OBJECTIVES:

I. Determine the effect of IFN-α-2b on tumor cell expression of CEA and MHC class I antigens in patients treated with this regimen.

II. Determine the immunologic effects of this regimen in these patients. III. Determine any objective anti-tumor responses that may occur in response to this regimen in these patients.

IV. Determine the time to tumor progression in patients treated with this regimen.

OUTLINE: This is a dose-escalation study of interferon alfa-2b (IFN-α-2b).

COURSE I: Patients receive recombinant vaccinia-CEA(6D)-TRICOM vaccine subcutaneously (SC) on day 1. Patients also receive sargramostim (GM-CSF) SC on days 1-4 and IFN-α-2b* SC on days 9, 11, and 13.

COURSES II-IV: Patients receive recombinant fowlpox-CEA(6D)-TRICOM vaccine SC on day 1. Patients also receive GM-CSF as in course 1 and IFN-α-2b* SC on days 1, 3, and 5.

NOTE: *The initial cohort of 6 patients does not receive IFN-α-2b.

Treatment repeats every 28 days for 4 courses in the absence of disease progression or unacceptable toxicity. After 4 courses, patients who do not have progressive disease or unacceptable toxicity may receive recombinant fowlpox-CEA (6D)-TRICOM vaccine, GM-CSF, and IFN-α-2b every 28 days for 2 more courses and then every 3 months for up to 2 years.

Cohorts of 3-6 patients receive escalating doses of IFN-α-2b until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity. Six additional patients are treated at the MTD; these patients must be HLA-A2 positive.

After completion of study treatment, patients are followed monthly for 4 months and then every 6-12 months for up to 15 years.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed carcinoembryonic antigen (CEA)-expressing carcinoma

  * Metastatic or locally advanced disease
* Tumor accessible for biopsy
* Must have received ≥ 1 prior systemic regimen for metastatic disease
* No known brain metastases
* Performance status - ECOG 0-2
* Performance status - Karnofsky 60-100%
* More than 6 months
* Absolute neutrophil count ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3
* Bilirubin ≤ 2.0 times upper limit of normal (ULN)
* AST and ALT ≤ 4.0 times ULN
* Hepatitis B negative
* Hepatitis C negative
* Creatinine ≤ 1.96 mg/dL
* Creatinine clearance > 50 mL/min
* No persistent proteinuria
* Protein < 1,000 mg by 24-hour urine collection
* No urinary sediment abnormalities
* No symptomatic congestive heart failure
* No unstable angina pectoris
* No cardiac arrhythmia
* No clinically significant cardiomyopathy requiring treatment
* No impaired function (i.e., ejection fraction < 50%) for patients who have not had prior vaccine and are asymptomatic
* HIV negative
* No ongoing or active infection
* No history of allergic reaction to eggs or egg products
* No history of allergy or untoward reaction to prior vaccinia vaccination (e.g., smallpox immunization) or to any of its components
* No history of or active eczema or other eczematoid skin disorders
* No atopic dermatitis
* No other acute, chronic, or exfoliative skin conditions, including any of the following:

  * Burns
  * Impetigo
  * Varicella zoster
  * Severe acne
  * Other open wounds or rashes
* No immunocompromised condition
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for ≥ 3 months after completion of study treatment

  * No sexual contact for 3 weeks after each vaccination treatment
* Must be willing to undergo tumor biopsy
* No psychiatric illness or social situation that would preclude study compliance
* No life-threatening illness
* No other active malignancy within the past 2 years except nonmelanoma skin cancer or superficial bladder or cervical lesions treated with surgical resection
* No other uncontrolled illness
* Must be able to avoid close household contact with the following individuals for ≥ 3 weeks after vaccinia vaccination:

  * Pregnant or nursing women
  * Children under 5 years of age
  * Individuals who are immunodeficient or immunosuppressed by disease or therapy (including HIV infection)
  * Individuals with the following conditions:

    * History of or active eczema or other eczematoid skin disorders
    * Atopic dermatitis
    * Other acute, chronic, or exfoliative skin conditions (e.g., burns, impetigo, varicella zoster, severe acne, or other open rashes or wounds)
* No concurrent influenza vaccine
* More than 4 weeks since prior chemotherapy (6 weeks for nitrosoureas or mitomycin) and recovered
* No concurrent steroid therapy, except topical or inhaled steroids
* No concurrent steroid eye drops
* More than 4 weeks since prior radiotherapy and recovered
* More than 4 weeks since prior surgery and recovered
* No prior splenectomy
* No other concurrent investigational agents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2005-06; Primary Completion 2013-01 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
MTD of IFN-alpha-2b, defined as the dose level one level beneath that dose at which 2 or more of 6 patients showed DLT, graded according to NCI CTCAE version 4.0 | Up to 112 days

SECONDARY OUTCOMES:
Incidence of adverse events, graded according to NCI CTCAE version 4.0 | Up to 15 years
  All patients will be evaluable for toxicity from the time of their first treatment with rF-CEA(6D)TRICOM and rV-CEA(6D)TRICOM.
Response to treatment, evaluated using the new international criteria proposed by the RECIST Committee | Up to 15 years
  Each patient will be assigned one of the following categories: 1) complete response, 2) partial response, 3) stable disease, 4) progressive disease, 5) early death from malignant disease, 6) early death from toxicity, 7) early death because of other cause, or 9) unknown (not assessable, insufficient data). Patients in response categories 4-9 should be considered as failing to respond to treatment (disease progression).

CONTACTS AND LOCATIONS:
Overall Officials: William Carson, Principal Investigator — Ohio State University Comprehensive Cancer Center
Locations (1):
- Ohio State University Comprehensive Cancer Center, Columbus, Ohio, United States